CLINICAL TRIAL: NCT03166059
Title: Prospective, Single Arm, Study to Assess the Safety and Performance of the CaveoVasc® Thrombolysis Protection System, for Femoral Artery Access and Protection in Patients Treated With Thrombolysis for Limb Ischemia
Brief Title: CaveoVasc Thrombolysis Protection System, Access Protection Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CaveoMed GmbH (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Caveomed-2017-05
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-05

CONDITIONS: Thrombolysis
Keywords: Catheter directed thrombolysis (CDT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): CaveoVasc® Thrombolysis Protection System
  Interventions: Device: CaveoVasc® Thrombolysis Protection System

INTERVENTIONS:
Device: CaveoVasc® Thrombolysis Protection System — CaveoVasc® Thrombolysis Protection System for Femoral Artery Access and Protection in Patients Treated with Thrombolysis for Limb Ischemia

SUMMARY:
The CaveoVasc Thrombolysis Protection System is intended to aid sheath access and reduce bleeding complications during catheter directed thrombolysis (CDT) in the treatment of limb ischemia. This device has been designed to protect the puncture site by stabilizing the CDT sheath with the double-balloons that are part of the CaveoVasc system. Also the device is designed to reduce bleeding at the puncture site during CDT.

This study is designed to assess the safety and performance of the CaveoVasc Thrombolysis Protection System in twenty patients with limb ischemia undergoing treatment with CDT.

DETAILED DESCRIPTION:
Catheter directed thrombolysis (CDT) is a non-surgical option for many patients, which involves the insertion of an infusion catheter (via the femoral artery) into the thrombus allowing for slow delivery of a pharmacological thrombolytic agent. Insertion of the infusion catheter is performed in the catheterization laboratory. The patient is usually then transferred to the intensive care unit, with delivery catheter in place and the infusion running for at least 24 hours.

The major complications reported with CDT include major and minor bleeding, and complications secondary to early termination of the CDT due to access site bleeding.

CaveoMed developed the CaveoVasc® Thrombolysis Protection System, a vascular access protection device intended for use in thrombolysis procedures. Its function is to facilitate sheath access, and minimize risks of access site bleeding complications during lengthy catheter-directed thrombolysis procedures. Pressure balloons inflated outside the artery maintain a good seal throughout thrombolysis, which typically lasts up to 24 hours. The thrombolysis catheter is then removed, and hemostasis at the site is managed per the hospital's standard.

The CaveoVasc® Thrombolysis Protection System design has important advantages for use during CDT procedures (which require long catheter dwell times). The system is intended to protect from intra-procedural bleeding at the arterial access site, which currently remains a major problem for patients with critical limb ischemia undergoing CDT treatment. This protection would lower the rate of bleeding events, and increase the rate of completed intended therapy, without interruption of the CDT treatment due to bleeding complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years
* Diagnosis of limb ischemia requiring CDT
* Patient understands and signs the study specific written informed consent form

Exclusion Criteria:

* Patients who are currently participating in another clinical trial of an investigational drug or device that has not concluded the follow-up period
* Patients who cannot adhere to or complete the investigational protocol for any reason
* Inability to provide informed consent or to comply with study assessments (e.g. due to cognitive impairment or geographic distance)
* Patients with bleeding disorders such as thrombocytopenia (platelet count<100,000/mm3), hemophilia, von Willebrand's disease or anemia (Hgb <10g/ dL, Hct < 30%)
* Patients who need a puncture needle longer than 8 cm due to morbid obesity
* Patients who are cachectic and do not have enough subcutaneous tissue/fat to accommodate the CaveoMed device (the two balloons, with 2 ml of contrast-enriched saline in each ballon)
* Patients who are pregnant or lactating
* Patients with documented INR > 1.5 or patients currently receiving glycoprotein IIb/IIIa platelet inhibitors, unless the glycoprotein IIb/IIIa platelet inhibitor is given as a bolus prior to the CDT as part of the institution's standard of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Rate of all major bleeds from the start of the CDT procedure to the end of the CDT procedure | Start of the CDT procedure to the end of the CDT procedure (usually less than 48 hours)
  BARC type > 3, as follows:
  Type 3 Type 3a Overt bleeding plus hemoglobin drop of 3 to <5 g/dL* (provided hemoglobin drop is related to bleed). Any transfusion with overt bleeding.
  Type 3b Overt bleeding plus hemoglobin drop >5 g/dL* (provided hemoglobin drop is related to bleed), cardiac tamponade, bleeding requiring surgical intervention for control (excluding dental/nasal/skin/hemorrhoid), bleeding requiring intravenous vasoactive agents.
  Type 3c Intracranial hemorrhage (does not include microbleeds or hemorrhagic transformation, does include intraspinal), subcategories confirmed by autopsy or imaging or lumbar puncture, intraocular bleed compromising vision.
  (Type 4: CABG-related bleeding is not applicable for this study) Type 5: fatal bleeding Type 5a Probable fatal bleeding; no autopsy or imaging confirmation but clinically suspicious Type 5b Definite fatal bleeding; overt bleeding or autopsy or imaging confirmation.
Duration of CDT procedure | Start of the CDT procedure to the end of the CDT procedure (usually less than 48 hours)
  Hours

SECONDARY OUTCOMES:
Adverse Events at Discharge | From consent to discharge (usually less than 48 hours from start of procedure)
  Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.
Adverse Events at 30 days | At 30 follow-up visit
  Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.
CDT without early interruption due to access site complication | Start to end of CDT procedure (usually less than 48 hours from start of procedure)
  Rate
Successful thrombolysis | Start to end of CDT procedure (usually less than 48 hours from start of procedure)
  Rate of successful thrombolysis without bleeding complication
Pain at access site | Start to end of lysis medication (usually less than 48 hours from start of procedure)
  verbal pain scale (0 to 10), at start of CDT (time when infusion of lysis medication started), after 6 hours of start of CDT, and at the end of the CDT treatment (time when infusion of lysis medication has stopped)

IPD SHARING:
Plan to Share IPD: No